CLINICAL TRIAL: NCT00714519
Title: A Phase II Feasibility Study of Xenaderm® Ointment Exploring Design Issues for Phase III Efficacy in Partial-Thickness Wounds
Brief Title: Feasibility Study of the Execution of an Efficacy Trial in the Nursing Home Setting
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to the inability to enroll subjects. No subjects were or ever will be enrolled into this study.
Sponsor: Healthpoint (Industry)
Responsible Party: Herbert Slade, MD/Chief Medical Officer, Healthpoint
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 011-101-09-032
Record Dates: First submitted 2008-07-10; First posted 2008-07-14 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Partial Thickness Wounds
Keywords: Xenaderm; partial; thickness; wounds; Nursing Homes
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Xenaderm® Ointment
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Xenaderm® Ointment — Topical, BID or as needed
  Other Names: Placebo Comparator
  Arms: 1
Drug: Placebo Comparator — Topical, BID or as needed
  Other Names: Xenaderm® Ointment
  Arms: 2

SUMMARY:
This study will assess if a clinical trial regarding healing of partial thickness wounds can be executed in nursing homes.

DETAILED DESCRIPTION:
This study will test the efficacy of Xenaderm® vs. vehicle on the healing of partial thickness wounds caused by pressure, moisture and friction.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent, which consists of reading, signing and dating the informed consent document after the Investigator, sub-Investigator or other designated study staff member has explained the study procedures, risks, and contact information. If the subject is unable to read or sign the informed consent, or unable to comprehend the information provided in the consent process, a legal guardian, decision making proxy, or next of kin must provide written consent, and if possible, subject must verbally assent to receiving an experimental treatment for their wound.
2. Are at least 18 years of age.
3. Are expected to remain in the Nursing Home for the duration of the study (22 days).
4. Have one or more partial-thickness wounds (including wounds with excoriation, erosion or denuded skin, or ulceration to subcutaneous fat, but with no fascia, muscle, tendon or bone visible) on the trunk or proximal extremity (arm above the elbow, leg above the knee) which

   * have been present for at least 2 days but less than 6 weeks;
   * measure greater than or equal to 2 and less than or equal to40 cm2 in total denuded area; and,
   * are connected by areas of erythema (for multiple wounds).
5. Are capable of maintaining an adequate nutritional intake during the study.
6. Are in an acceptable state of health and nutrition with pre-albumin levels of greater than or equal to 15 mg/dl (0.015g/l), serum albumin greater than or equal to 3.0 g/dl (30g/l), alkaline phosphatase greater than or equal to the lower limit of normal, and have no abnormal laboratory values that, in the opinion of the Medical Supervisor, place the subject at risk for the study.

Exclusion Criteria:

1. Have more than 64 cm2 of total denuded wound area, including target and non-target wounds.
2. Have a full-thickness wound within 4 cm of any target wound.
3. Have clinical evidence of bacterial or fungal infection of the target wound.
4. Have target wound(s) that involves tunneling, sinus tracks, shear injury, arterial occlusive disease or bony prominence or joint with the exception that target wounds may be over dorsal spinous processes, coccyx, ischial tuberosities or sacroiliac joints (but may not be full thickness).
5. Are moribund, or has a severe burn, immunodeficiency disorder, hematologic disorder, metastatic malignancy or uncontrolled diabetes mellitus.
6. Are known to have acrodermatitis enteropathica (zinc deficiency).
7. Are being treated with systemic steroids, immunosuppressive agents, radiation or chemotherapy.
8. Have been treated with enzymatic debridement to the target wound(s) within 2 days prior to enrollment.
9. Have a known sensitivity to ingredients of Xenaderm Ointment.
10. Are using or have used another investigational agent (not including devices such as hearing aids, pace makers, etc.) within 30 days prior to Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Complete Wound Closure | 21 days

SECONDARY OUTCOMES:
Adverse Events | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Herbert B Slade, MD, Study Chair — Healthpoint; Innes Cargill, PhD, Study Director — Healthpoint